CLINICAL TRIAL: NCT00256672
Title: Effectiveness of Full-Time Prophylactic Bracing at Preventing or Delaying Curve Progression in Paralytic Scoliosis Secondary to Spinal Cord Injury in the Growing Child: Randomized Trial
Brief Title: Effectiveness of Bracing in Preventing Scoliosis in Children With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Craig McDonald, MD, principal investigator, Shriners Hospital for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9155-200513332
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Scoliosis
Keywords: Spinal Cord Injury; TLSO brace; Spine curvature; Child; Effectiveness of bracing
MeSH Terms: conditions — Scoliosis; Spinal Cord Injuries; Spinal Curvatures

ARMS (2):
- 1 (Active Comparator): High-dose Thoraco-Lumbar-Sacral Orthoses wear (>23hrs/day) will be compared to low-dose Thoraco-Lumbar-Sacral Orthoses wear (12hrs/day)
  Interventions: Device: Thoraco-Lumbar-Sacral-Orthoses (TLSO) / Flex-Foam
- 2 (Active Comparator): Low-dose Thoraco-Lumbar-Sacral-Orthoses wear (12hrs/day)
  Interventions: Device: Thoraco-Lumbar-Sacral-Orthoses (TLSO) / Flex-Foam

INTERVENTIONS:
Device: Thoraco-Lumbar-Sacral-Orthoses (TLSO) / Flex-Foam — TLSO back brace, Flex-Foam (Posterior Opening)

SUMMARY:
The purpose of this study is to determine whether full-time high dose prophylactic bracing (23 hours or more per day) is more effective than low dose bracing (12 hours or less per day) in preventing or delaying spinal curve progression in children with scoliosis after spinal cord injury.

DETAILED DESCRIPTION:
This is a randomized control trial to determine the effectiveness of high dose bracing (≥ 23 hours per day) and low dose bracing (≤ 12 hours per day) in skeletally immature children with Spinal Cord Injury. Subjects will be randomized into either a prophylactic high dose-bracing group (≥ 23 hours per day) or low dose-bracing group (≤ 12 hours per day). Subjects will be stratified by age (younger than age 10 and older than age 10), and curve severity (< 20 degrees and 20-40 degrees) using a matching random blocks design.

ELIGIBILITY:
Inclusion Criteria:

1. Children with C5 to L2 SCI.
2. ASIA impairment levels A, B, or C.
3. Age greater than 5 up to one year before end of growth (14 in girls, 16 in boys)
4. A single structural curve <40 degrees or a double curve <40 degrees where the largest compensatory curve is <25 degrees on bending film.
5. Children at risk for Paralytic Scoliosis
6. Ability to follow simple instructions.

Exclusion Criteria:

1. Curve magnitude >40 degrees, pressure sores over the trunk.
2. Inability to tolerate TLSO wears.
3. Structural compensatory curves of 25 degrees or greater (double structural curves).
4. Severe Traumatic Brain Injury, TBI (8 and below on Glasgow Coma Scale).
5. Cognitive Impairment
6. Less than 6 months from date of injury

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
X-rays (at the time of consent and every 6 months for 5 years) to determine degree of scoliosis. | 5 years
Timed Motor Assessment (at the time of consent and once a year for 5 years) to measure functional ability in daily life activities including putting on sweat pants, T-Shirt, transferring from wheelchair to bed, etc. | 5 years
Reachable Workspace Assessment (at the time of consent and once a year for 5 years): performing functional tasks including reaching for the floor, overhead, and every 20-degree radius in between. | 5 years
Global Measures (at the time of consent and every 6 months for 5 years): Four different questionnaires to monitor function, satisfaction, and quality of life. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig M McDonald, MD, Principal Investigator — Shriners Hospital for Children, Northern California; Randal R Betz, MD, Principal Investigator — Shriners Hospital for Children, Philadelphia; Lawrence Vogel, MD, Principal Investigator — Shriners Hospital for Children, Chicago
Locations (3):
- United States (3):
  - Shriners Hospital for Children - Northern California, Sacramento, California
  - Shriners Hospital for Children - Chicago, Chicago, Illinois
  - Shriners Hospital for Children - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Rab G, Petuskey K, Bagley A. A method for determination of upper extremity kinematics. Gait Posture. 2002 Apr;15(2):113-9. doi: 10.1016/s0966-6362(01)00155-2. PMID 11869904
- [Background] Kukke SN, Triolo RJ. The effects of trunk stimulation on bimanual seated workspace. IEEE Trans Neural Syst Rehabil Eng. 2004 Jun;12(2):177-85. doi: 10.1109/TNSRE.2004.827222. PMID 15218932
- [Background] Palmieri TL, Petuskey K, Bagley A, Takashiba S, Greenhalgh DG, Rab GT. Alterations in functional movement after axillary burn scar contracture: a motion analysis study. J Burn Care Rehabil. 2003 Mar-Apr;24(2):104-8. doi: 10.1097/01.BCR.0000054170.62555.09. PMID 12626930
- [Background] Betz RR & Mulcahey MJ. Spinal Cord Injury Rehabilitation, In: The Pediatric Spine: Principles and Practice, S.L. Weinstein (eds). New York: Raven press, 1994.
- [Background] Brown JC, Zeller JL, Swank SM, Furumasu J, Warath SL. Surgical and functional results of spine fusion in spinal muscular atrophy. Spine (Phila Pa 1976). 1989 Jul;14(7):763-70. doi: 10.1097/00007632-198907000-00020. PMID 2772729
- [Background] Campbell J, Bonnett C. Spinal cord injury in children. Clin Orthop Relat Res. 1975 Oct;(112):114-23. PMID 1192626
- [Background] Dearolf WW 3rd, Betz RR, Vogel LC, Levin J, Clancy M, Steel HH. Scoliosis in pediatric spinal cord-injured patients. J Pediatr Orthop. 1990 Mar-Apr;10(2):214-8. PMID 2312704
- [Background] Lou E, Raso JV, Hill DL, Durdle NG, Mahood JK, Moreau MJ. The daily force pattern of spinal orthoses in subjects with adolescent idiopathic scoliosis. Prosthet Orthot Int. 2002 Apr;26(1):58-63. doi: 10.1080/03093640208726622. PMID 12043927
- [Background] Lancourt JE, Dickson JH, Carter RE. Paralytic spinal deformity following traumatic spinal-cord injury in children and adolescents. J Bone Joint Surg Am. 1981 Jan;63(1):47-53. PMID 7451526
- [Background] Lou E, Raso J, Hill D, Durdle N, Mahood J, Moreau M. Brace monitoring system for the treatment of scoliosis. Stud Health Technol Inform. 2002;88:218-21. PMID 15456036
- [Background] DiRaimondo CV, Green NE. Brace-wear compliance in patients with adolescent idiopathic scoliosis. J Pediatr Orthop. 1988 Mar-Apr;8(2):143-6. PMID 3350947
- [Background] Gurnham RB. Adolescent compliance with spinal brace wear. Orthop Nurs. 1983 Nov-Dec;2(6):13-7. doi: 10.1097/00006416-198311000-00003. No abstract available. PMID 6562445
- [Background] Havey R, Gavin T, Patwardhan A, Pawelczak S, Ibrahim K, Andersson GB, Lavender S. A reliable and accurate method for measuring orthosis wearing time. Spine (Phila Pa 1976). 2002 Jan 15;27(2):211-4. doi: 10.1097/00007632-200201150-00018. PMID 11805670
- [Background] Lindeman M, Behm K. Cognitive strategies and self-esteem as predictors of brace-wear noncompliance in patients with idiopathic scoliosis and kyphosis. J Pediatr Orthop. 1999 Jul-Aug;19(4):493-9. doi: 10.1097/00004694-199907000-00013. PMID 10412999
- [Background] Lou E, Durdle NG, Raso VJ, Hill DL: A Load Compliance Monitor System for the Treatment of Scoliosis. Proceedings of IEEE Canadian Conference on Electrical and Computer Engineering, Edmonton, Canada pp. 1501-1505, 1999.
- [Background] Mayfield JK. Severe spine deformity in myelodysplasia and sacral agenesis: an aggressive surgical approach. Spine (Phila Pa 1976). 1981 Sep-Oct;6(5):498-509. doi: 10.1097/00007632-198109000-00013. PMID 7302685
- [Background] Mayfield JK, Erkkila JC, Winter RB. Spine deformity subsequent to acquired childhood spinal cord injury. J Bone Joint Surg Am. 1981 Dec;63(9):1401-11. PMID 7320032
- [Background] Vandal S, Rivard CH, Bradet R. Measuring the compliance behavior of adolescents wearing orthopedic braces. Issues Compr Pediatr Nurs. 1999 Apr-Sep;22(2-3):59-73. doi: 10.1080/014608699265293. PMID 10786513
- [Background] Chafetz R, McDonald C, Mulcahey MJ, Betz R, Anderson C, Vogel L, Gaughan JP, Martin S, O'Dell MA, Flanagan A. Timed motor test for wheelchair users: initial development and application in children with spinal cord injury. J Spinal Cord Med. 2004;27 Suppl 1:S38-43. doi: 10.1080/10790268.2004.11753783. PMID 15503701
- [Background] Anderson C A, Vogel L C, Klaas SJ, Lubicky J P, Long-term outcomes and life satisfaction in pediatric spinal cord injury: a model for children with chronic disabilities. (Presented at the annual meeting of the American Academy of Cerebral Palsy and Developmental Medicine 1997). Dev. Med. Child Neurol. 1997; 39 (Suppl 75): 21.
- [Background] Bonaroti D, Akers JM, Smith BT, Mulcahey MJ, Betz RR. Comparison of functional electrical stimulation to long leg braces for upright mobility for children with complete thoracic level spinal injuries. Arch Phys Med Rehabil. 1999 Sep;80(9):1047-53. doi: 10.1016/s0003-9993(99)90059-x. PMID 10489007
- [Background] Bridwell KH, Baldus C, Iffrig TM, Lenke LG, Blanke K. Process measures and patient/parent evaluation of surgical management of spinal deformities in patients with progressive flaccid neuromuscular scoliosis (Duchenne's muscular dystrophy and spinal muscular atrophy). Spine (Phila Pa 1976). 1999 Jul 1;24(13):1300-9. doi: 10.1097/00007632-199907010-00006. PMID 10404571
- [Background] Daltroy LH, Liang MH, Fossel AH, Goldberg MJ. The POSNA pediatric musculoskeletal functional health questionnaire: report on reliability, validity, and sensitivity to change. Pediatric Outcomes Instrument Development Group. Pediatric Orthopaedic Society of North America. J Pediatr Orthop. 1998 Sep-Oct;18(5):561-71. doi: 10.1097/00004694-199809000-00001. PMID 9746401
- [Background] Deutsch A, Braun S, Granger CV. The Functional Independence Measure and the Functional Independence Measure for Children: ten years of development. Crit Rev Med Rehab 1996; 8:267-281.
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Law M, Polatajko H, Pollock N, McColl MA, Carswell A, Baptiste S. Pilot testing of the Canadian Occupational Performance Measure: clinical and measurement issues. Can J Occup Ther. 1994 Oct;61(4):191-7. doi: 10.1177/000841749406100403. PMID 10137673
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- See also: Official website for Shriners Hospitals for Children, a network of 22 hospitals that provide expert, no-cost orthopaedic and burn care to children under 18 — http://www.shrinershq.org